CLINICAL TRIAL: NCT06126146
Title: Patient-reported Real-world Experience of Risankizumab On-body Injector (OBI) for the Treatment of Crohn's Disease in the UK: a Before-and-after Survey of Participants Among Patients That Transition From Maintenance Treatment (360 mg Applied by 4x90 mg PFS) Within the Early Access to Medicine Scheme / Pre-Approval Access Schemes to OBI
Brief Title: An Observational Study to Assess Participant-Reported Real-World Experience of Risankizumab On-body Injector (OBI) for the Treatment of Crohn's Disease in Adult Participants in the United Kingdom (UK)
Acronym: COMMODUS
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P24-171
Record Dates: First submitted 2023-11-07; First posted 2023-11-13 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2024-05

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease; Risankizumab; Skyrizi
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Risankizumab: Participants will receive risankizumab on-body injector (OBI) as prescribed by their physician according to local label.

SUMMARY:
Crohn's Disease (CD) is a chronic condition that causes inflammation of the gastrointestinal tract or gut. This study will assess real-world, adult participant experience of self-injection with the risankizumab OBI.

Risankizumab is an approved drug for the treatment of CD in adults. Approximately 80 participants who are prescribed risankizumab by their doctors and are transitioning from the pre-filled syringe (PFS) to the use of OBI will be enrolled in this study in the United Kingdom (UK).

Participants will receive risankizumab OBI as prescribed by their physician according to their routine clinical practice and local label. Participants will be followed for up to 6 months.

There is expected to be no additional burden for participants in this trial. Study visits may be conducted on-site, at home, or virtually as per standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Eligible for and received risankizumab for maintenance treatment of Crohn's Disease (CD) through United Kingdom (UK) Early Access to Medicines Scheme (EAMS)/Pre-Approval Access (PAA) schemes
* The decision to treat with risankizumab was made independently, in line with usual clinical practice, marketing authorisation and prior to enrolment in the study
* Exits UK EAMS/PAA and switches from risankizumab pre-filled syringe (PFS) to on-body injector (OBI)
* Can physically self-administer risankizumab OBI without carer assistance
* Can read and understand English
* Willing and able to provide voluntary informed consent
* Able and willing to participate in this study.

Exclusion Criteria:

N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults who received risankizumab for maintenance treatment of CD through United Kingdom (UK) Early Access to Medicines Scheme (EAMS)/Pre-Approval Access (PAA) schemes who are due to switch from risankizumab pre-filled syringe (PFS) to use of on-body injector (OBI).
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2023-10-26 (Actual); Primary Completion 2024-05-16 (Actual); Study Completion 2024-05-16 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Individual Item Score in Response to Q18 "Overall, how satisfied are you with your current way of taking your medication (self injection)?" in Post-Injection Self-Injection Assessment Questionnaire (SIAQ) | Baseline up to approximately 6 months
  SIAQ evaluations consist of the PRE module, which is self-completed immediately before the first OBI self-injection at baseline, and the POST module, which is self-completed following injections.
  Participants rate each item of the SIAQ. The ratings are later transformed to scores ranging from 0 (worst experience) to 10 (best experience). The domain score is the mean of the item scores included in the domain. Domain scores are calculated only if at least half of the domain items are completed. Item and domain scores from the PRE module are compared with the corresponding item and domain scores from the POST modules.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (5):
- United Kingdom (5):
  - University Hospital Southampton NHS Foundation Trust /ID# 258989, Southampton, Hampshire
  - Guys and St Thomas NHS Foundation Trust /ID# 258986, London, London, City of
  - NHS Lothian /ID# 260901, Edinburgh
  - The Royal London Hospital /ID# 259047, London
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust /ID# 260902, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Clinical Study Report Synopsis — https://www.abbvieclinicaltrials.com/study/?id=P24-171#additional-resources-section